CLINICAL TRIAL: NCT01742650
Title: Screw Versus Tightrope Syndesmotic Injury Fixation in Weber C Ankle Fractures. A Prospective Randomized Study.
Brief Title: Screw Versus Tightrope Syndesmotic Injury Fixation in Weber C Ankle Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Harri Pakarinen, MD, PhD, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OYS-7-2009
Record Dates: First submitted 2012-06-12; First posted 2012-12-05 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Trauma
Keywords: ankle; fracture; syndesmosis;
MeSH Terms: conditions — Wounds and Injuries; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Screw fixation (Active Comparator): 3,5mm fully threaded cortical screw transfixation of syndesmosis
  Interventions: Procedure: Screw fixation
- TightRope (Active Comparator): TightRope transfixation of syndesmosis
  Interventions: Procedure: TightRope

INTERVENTIONS:
Procedure: Screw fixation — 3,5mm fully threaded cortical screw transfixation of syndesmosis
  Arms: Screw fixation
Procedure: TightRope — TightRope transfixation of syndesmosis
  Other Names: Tightrope Arthrex
  Arms: TightRope

SUMMARY:
The aim of our study is to compare two different syndesmosis transfixation methods in AO/OTA Weber C ankle fractures. Our hypothesis is that 50% of screw fixed fibulas but only 5% of suture-button fixed fibulas are in malposition. All skeletally mature patients (16 years or older) with AO/OTA Weber C type fractures operated within a week after trauma are consecutively included into the study. The tibiofibular transfixation is randomly performed either by a 3,5 mm tricortical screw or a suture-button (TightRope). Malposition of the tibiofibular joint is assessed in an intraoperative computed tomography. Clinical outcome is assessed by using Olerud-Molander, RAND ja 36-Item Healt Survey after 1-year from the injury.

DETAILED DESCRIPTION:
The aim of our study is to compare two different syndesmosis transfixation methods in AO/OTA Weber C ankle fractures. Screw fixation is widely and mostly used transfixation but suture-button is also shown to be a biomechanically stable and probably more physiologic transfication method. It is shown that even 50 % of the syndesmosis srews and thus fibulas are in malposition. With more physiologic suture-button transfixation this malposition is thought to be less commmon. There is no studies comparing screw and suture-button syndesmosis transfixation methods in AO/OTA Weber C ankle fracture patients.

Our hypothesis is that 50% of screw fixed fibulas but only 5% of suture-button fixed fibulas are in malposition assessed in the intraoperative computed tomography. Malposition is assessed to present if difference between fractured and non-fractured side is at least 2 mm in the tibiofibular joint. Thus, the sample size is assessed to be 19 patients per group (alpha=0.05, Beta=0.2, 20% drop out).

All skeletally mature patients (16 years or older) with AO/OTA Weber C type fractures operated within a week after trauma are included into the study. Exclusion criteria are previous ankle fracture, concomitant tibial fracture, diabetes with peripheral neuropathy, pathological fracture or inadequate co-operation.

After bony fixation the tibiofibular transfixation is randomly performed either by a 3,5 mm tricortical screw or a suture-button (TightRope). An intraoperative computed tomography is imaged from the both ankles of all patients. The operation is continued with six weeks casting without weight-bearing.

Clinical outcome was assessed using the Olerud-Molander scoring system, RAND 36-Item Health Survey, and Visual Analogue Scale (VAS) to measure pain and function after a minimum 1-year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* AO/OTA Weber C ankle fracture, operation within 7 days from the injury

Exclusion Criteria:

* Bilateral or previous ankle fracture, tibial shaft fracture, diabetes wiht polyneuropathy, inadequate co-operation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Malreduction of the tibiofibular joint in the intraoperative computed tomography | 2 years
  Malreduction in the tibiofibular joint is assessed post op from the intraoperative computed tomography. Both ankles are imaged and difference at least 2 mm is assessed to be significant

SECONDARY OUTCOMES:
Clinical outcome one year after the injury | 2 year
  Clinical outcome was assessed using the Olerud-Molander scoring system, RAND 36-Item Health Survey, and Visual Analogue Scale (VAS) to measure pain and function after a minimum 2-year of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Tero HJ Kortekangas, MD, Principal Investigator — Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kortekangas T, Savola O, Flinkkila T, Lepojarvi S, Nortunen S, Ohtonen P, Katisko J, Pakarinen H. A prospective randomised study comparing TightRope and syndesmotic screw fixation for accuracy and maintenance of syndesmotic reduction assessed with bilateral computed tomography. Injury. 2015;46(6):1119-26. doi: 10.1016/j.injury.2015.02.004. Epub 2015 Feb 21. PMID 25769201